CLINICAL TRIAL: NCT04560829
Title: Additive Value of Physiology Coronary in Clinical Practice
Acronym: PRINCIPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.294; 2020-A02325-34 (Other: ID RCB)
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Microvascular Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The important evidence of coronary microcirculation for the management of patients with coronary artery disease is only increasing. Thus, in recent years, a number of studies have shown that the demonstration of coronary microvascular disease (CMVD) contributes to cardiovascular morbidity and mortality increases independently of epicardial damage. This has been shown in stable coronary artery disease with screening for CMVD when there is no significant epicardial involvement and allowing the implementation of an adapted treatment then reducing the symptoms and improving the quality of life of our patients. (1). The prognostic nature of CMVD has also been identified in stable disease after coronary angioplasty (2) but also in patients with infarcts reperfused by coronary angioplasty (3).

The complete exploration of the epicardial and microvascular coronary vascularization is grouped under the name of the subspecialty: coronary physiology. Thus, an internationally recognized algorithm for exploring coronary physiology has been published (4).

However, this algorithm is still little followed. The PRINCIPE registry aims to assess the prevalence of CMVD with the use of a standardized algorithm for exploring coronary physiology by coronary angiography in our center in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age
* Having a coronary angiography
* Presenting in pain or having performed a positive ischemia test
* Affiliated with social security
* Non-opposition to participation

Exclusion Criteria:

* Adult patient protected by law (article L1121-8)
* Person deprived of liberty (article L1121-8)
* Pregnant woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing coronary artery assessment. Patients will be included in the study prospectively during the assessment with collection of the patient's non-objection during follow-ups.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Rate of CMVD defined by microcirculatory resistance index (IMR) > 25 | At inclusion

SECONDARY OUTCOMES:
Prevalence of macro and microvascular angina | At inclusion
  Macro and microvascular angina rate according to international angiographic diagnostic criteria
Correlation between coronary physiology parameters and imaging data | At inclusion
  Coronary angiography and coronary physiology parameters:% of epicardial stenosis, FFR, CFR, IMR
Correlation between coronary physiology parameters and imaging data | At inclusion
  SPEC parameters
Correlation between coronary physiology parameters and imaging data | At inclusion
  Cardiac echography parameters
Correlation between coronary physiology parameters and imaging data | At inclusion
  Stress cardiac echography parameters
Correlation between coronary physiology parameters and imaging data | At inclusion
  MRI parameters
Correlation between coronary physiology parameters and imaging data | At inclusion
  Cardiac CT parameters
Assessment of the symptoms of angina pectoris | 12 months
  Brief angina questionnaire
Compare the rate of peri-procedural myocardial distress | At inclusion
  Post PCI troponin rate
Evaluate medical consumption | 12 months
  Number of medical consultation
Evaluation of serious cardiovascular event rate | 12 months
  Cardiovascular event

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided